CLINICAL TRIAL: NCT05811156
Title: A Biopsychosocial Treatment Model for Exhaustion Due to Persistent Non-traumatic Stress, Administered Through a Multimodal Digital Intervention - A Pilot Study
Brief Title: A Biopsychosocial Treatment for Exhaustion Due to Persistent Non-traumatic Stress
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: PBM Sweden AB (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-06789-01
Record Dates: First submitted 2023-02-20; First posted 2023-04-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: Exhaustion Disorder; Clinical Burnout

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Hybrid Multimodal digital intervention — Multimodal digital intervention, including an internet-delivered CBT treatment based on a biopsychosocial exposure treatment, tailored explicitly for Exhaustion due to persistent non-traumatic stress.
  Other Names: Internet CBT

SUMMARY:
Currently, there are no established theoretical models for developing and maintaining Exhaustion due to persistent non-traumatic stress (ENTS). Therefore, the current pilot study aims to evaluate a Multimodal hybrid intervention built around an internet-delivered cognitive behavioral therapy based on a new biopsychosocial treatment model of ENTS.

DETAILED DESCRIPTION:
Since 2009 long term sick-leave rates due to mental disorders have been increasing in Sweden and are today the leading cause of long-term sick leave. Exhaustion due to persistent non-traumatic stress (ENTS) accounts for most of this increase. Unfortunately, despite several published treatment studies, no evidence-based treatments exist for ENTS, and little is still known about the focus of treatment.

Currently, there are no established theoretical models for the development and maintenance of ENTS. Many of the published clinical ENTS trials consist of long (6 months or more) Multimodal interventions (MMI) containing various medical, psychological, and physiotherapeutic methods with a low degree of understanding of what components are critical for treatment success. Even if ENTS patients participating in MMI report symptom improvements and work resumption, MMI is generally personnel intensive and challenging to administer. These factors increase the risk of extended healthcare lead times and obstruct treatment dissemination.

Considering the increasing sick-leave rates due to ENTS, there is an apparent need for more accessible treatments based on pronounced theoretical models focusing on specific change processes. Therefore, the current pilot study aims to evaluate a hybrid MMI built around an internet-delivered cognitive behavioral therapy based on a new biopsychosocial treatment model of ENTS.

Outcome measures will be collected before and after treatment and at three and six-month follow-ups. Weekly measurements of putative processes of change will also be collected. The current study aims to evaluate whether this more restricted and theoretically coherent hybrid MMI shows promising results before we test the treatment solely as a cognitive behavioral therapy via the internet in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Referred for Stress-induced exhaustion disorder (SED)
* Fulfilled the criteria for SED
* Scored > 5 on the Shirom-Melamed Burnout Questionnaire (a cut-off determined by the Health Care Services Stockholm County)
* Scored 19 > on Karolinska Exhaustion Disorder Scale
* In need of sick-leave due to SED d) access to internet

Exclusion Criteria:

* 100 % sick leave of more than one year
* abuse of alcohol or drugs
* participating in any other form of MMI
* severe depression, moderate/high risk of suicide, psychosis, or untreated PTSD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SED who are accepted to treatment for a Multimodal digital intervention within a specialized healthcare initiative called "The healthcare choice for treatment of longstanding pain with or without comorbidity, and SED."
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Karolinska Exhaustion Disorder Scale | Baseline measurement, weekly (up to 12 weeks) change during from treatment baseline to immediately after treatment, change between immediately after treatment and 3 months follow-up, change between 3 months follow up and 6 months follow-up
  Measures symptoms of Exhaustion. It is specifically tailored to measure symptoms from the Swedish diagnosis of Stress-induced exhaustion disorder.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline, change between baseline and immediately after treatment, change between immediately after treatment and 6 months follow-up
  Measure of depression and anxiety
Flourishing scale | Baseline, change between baseline and immediately after treatment, change between immediately after treatment and 6 months follow-up
  brief 8-item summary measure of the respondent's self-perceived success in important areas such as relationships, self-esteem, purpose, and optimism
The current percentage of working time and sick-leave | Baseline, change between baseline and immediately after treatment, change between immediately after treatment and 6 months follow-up
  Rated by independent rater through telephone interview
WHO Disability Assessment Schedule 2.0-12 (Rated by independent rater) | Baseline, change between baseline and immediately after treatment, change between immediately after treatment and 6 months follow-up
  Measures difficulties due to health conditions
Client satisfaction Questionnaire- 8 | immediately after treatment
  Measure of treatment satisfaction
Negative Effects Questionnaire | immediately after treatment
  Measures negative effects attributable to treatment

OTHER OUTCOMES:
Perfectionistic concerns, sub scale av Clinical Perfectionism Questionnaire | weekly (for up to 12 weeks) change during from treatment baseline to end of treatment,
  A measure of perfectionistic concerns, a putative process variable in treatment
Penn-state worry questionnaire-brief | weekly (for up to 12 weeks) change during from treatment baseline to end of treatment,
  A measure of pathological worry, a putative process variable in treatment
Psy-flex | weekly (for up to 12 weeks) change during from treatment baseline to end of treatment,
  A measure of psychological flexibility, a putative process variable in treatment
Insomnia severity index (3-item version) | weekly (for up to 12 weeks) change during from treatment baseline to end of treatment,
  A measure of psychological dimensions of insomnia, a putative process variable in treatment

CONTACTS AND LOCATIONS:
Locations (1):
- PBM Sweden AB Globen, Stockholm, Södermanland County, Sweden

IPD SHARING:
Plan to Share IPD: No